CLINICAL TRIAL: NCT02789631
Title: Relationship Between Musculoskeletal, Sensorimotor and Functional Factors and Nonspecific Chronic Neck Pain
Status: Completed | Type: Observational
Sponsor: University of Social Welfare and Rehabilitation Science (Other)
Responsible Party: Principal Investigator, Dr. L. Ghamkhar, PhD Candidate, University of Social Welfare and Rehabilitation Science
Other Study IDs: IR.USWR.REC.1394.224
Record Dates: First submitted 2016-04-22; First posted 2016-06-03 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- chronic neck pain: experiencing neck pain for at least 3 months in the last year
  Interventions: Other: assessment
- without neck pain (asymptomatic): no history of neck pain
  Interventions: Other: assessment

INTERVENTIONS:
Other: assessment

SUMMARY:
Several factors have been associated with neck pain. Controversy exists regarding the degree of association between some of these factors and neck pain. Information regarding the degree of association of each factor to neck pain is needed for effective prevention and appropriate treatment strategies. The aim of this study is to investigate the association among musculoskeletal, sensorimotor factors and functional disability and occurrence of chronic nonspecific neck pain.

ELIGIBILITY:
Inclusion Criteria:

* for subjects with neck pain: experiencing pain for at least 3 months in the last year, having pain score of 3 or more on visual analogue scale.
* for healthy subjects: no history of neck pain

Exclusion Criteria:

* history of cervical discopathy
* any surgery on neck
* traumatic neck injury
* any congenital disorders

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: subjects with and without neck pain
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2015-10; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
flexor and extensor cervical muscles holding time (second) | 2 years
cervical, back, lowback, upper limbs, lower limbs muscles and trunk maximal contraction force against resistance (N) | 2 years
head inclination angle, lumbar and thoracic angles in sagittal plane and thoracic angle in the coronal plane (degrees) | 2 years
pelvic inclination in the sagittal and coronal planes (degrees) | 2 years
cervical, back, low back, upper limbs, lower limbs and trunk range of motion in sagittal and coronal planes (degrees) | 2 years
cervical re-positioning error (degrees) | 2 years
the result of Dixhallpike test (positive or negative for vertigo and nystagmus) | 2 years
neck disability questionnaire score | 2 years
distance between T2 spinous process and spine of the scapula (cm) | 2 years
the difference between chest circumference at xiphoid process, axillary and umbliqus levels in the inhalation and exhalation phases of respiration (cm) | 2 years
the result of the Romberg test (seconds) | 2 years
the result of the upper cervical flexion with rotation test (positive/negative) | 2 years
the result of the Gaze test (positive/negative) | 2 years
pain reproduction test by the algometer at 2.5 kg pressure level (positive/negative) | 2 years
visual analogue scale score | 2 years

SECONDARY OUTCOMES:
Pearson correlation coefficient of the cervical muscles holding time with visual analogue scale score | 2 years
Pearson correlation coefficient of the cervical muscles holding time with neck disability index questionnaire score | 2 years
Pearson correlation coefficient of cervical, back, lowback, upper limbs, lower limbs muscles and trunk maximal contraction force against resistance with neck disability index questionnaire score | 2 years
Pearson correlation coefficient of cervical, back, lowback, upper limbs, lower limbs muscles and trunk maximal contraction force against resistance with visual analogue scale score | 2 years
Pearson correlation coefficient of head inclination angle, lumbar and thoracic angles in sagittal plane and thoracic angle in the coronal plane with visual analogue scale score | 2 years
Pearson correlation coefficient of head inclination angle, lumbar and thoracic angles in sagittal plane and thoracic angle in the coronal plane with neck disability index score | 2 years
Pearson correlation coefficient of pelvic inclination in the sagittal and coronal planes with neck disability index score | 2 years
Pearson correlation coefficient of pelvic inclination in the sagittal and coronal planes with visual analogue scale score | 2 years
Pearson correlation coefficient of cervical, back, low back, upper limbs, lower limbs and trunk range of motion in sagittal and coronal planes with neck disability index score | 2 years
Pearson correlation coefficient of cervical, back, low back, upper limbs, lower limbs and trunk range of motion in sagittal and coronal planes with visual analogue scale score | 2 years
Pearson correlation coefficient of the difference between chest circumference at xiphoid process, axillary and umbliqus levels in the inhalation and exhalation phases of respiration with visual analogue scale score | 2 years
Pearson correlation coefficient of the difference between chest circumference at xiphoid process, axillary and umbliqus levels in the inhalation and exhalation phases of respiration with neck disability index score | 2 years
Pearson correlation coefficient of distance between T2 spinous process and spine of the scapula with neck disability index score | 2 years
Pearson correlation coefficient of distance between T2 spinous process and spine of the scapula with visual analogue scale score | 2 years
Pearson correlation coefficient of cervical re-positioning error with visual analogue scale score | 2 years
Pearson correlation coefficient of cervical re-positioning error with neck disability index score | 2 years
Pearson correlation coefficient of Romberg test with neck disability index score | 2 years
Pearson correlation coefficient of Romberg test with visual analogue scale score | 2 years
Spearman correlation coefficient of pain reproduction test by the algometer at 2.5 kg pressure level with visual analogue scale score | 2 years
Spearman correlation coefficient of pain reproduction test by the algometer at 2.5 kg pressure level with neck disability index score | 2 years
Spearman correlation coefficient of the result of the upper cervical flexion with rotation test with neck disability index score | 2 years
Spearman correlation coefficient of the result of the upper cervical flexion with rotation test with visual analogue scale score | 2 years
Spearman correlation coefficient of the result of Dixhallpike test with visual analogue scale score | 2 years
Spearman correlation coefficient of the result of Dixhallpike test with neck disability index score | 2 years
Spearman correlation coefficient of the result of Gaze test with neck disability index score | 2 years
Spearman correlation coefficient of the result of Gaze test with visual analogue scale score | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Social Welfare and Rehabilitation Sciences, Tehran, Iran

REFERENCES:
- [Derived] Kahlaee AH, Ghamkhar L, Nourbakhsh MR, Arab AM. Strength and Range of Motion in the Contralateral Side to Pain and Pain-Free Regions in Unilateral Chronic Nonspecific Neck Pain Patients. Am J Phys Med Rehabil. 2020 Feb;99(2):133-141. doi: 10.1097/PHM.0000000000001298. PMID 31464752